CLINICAL TRIAL: NCT03897868
Title: A Muticenter, Randomized, Double-blind, Parallel, Phase 2 Study to Assess Dose-response Relationship of HCP1803 in Patients With Essential Hypertension
Brief Title: A Phase 2 Study to Assess Dose-response Relationship of HCP1803 in Patients With Essential Hypertension
Acronym: HM_APOLLO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-APOLLO-201
Record Dates: First submitted 2019-03-29; First posted 2019-04-01 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Experimental 1 (Experimental): HCP1803 High
  Interventions: Drug: HCP1803; Drug: Placebo
- Experimental 2 (Experimental): HCP1803 Middle
  Interventions: Drug: HCP1803; Drug: Placebo
- Experimental 3 (Experimental): HCP1803 Low
  Interventions: Drug: HCP1803; Drug: Placebo
- Active Comparator 1 (Active Comparator): HGP0904 High
  Interventions: Drug: Amlodipine
- Active Comparator 2 (Active Comparator): HGP0904 Low
  Interventions: Drug: Amlodipine; Drug: Placebo
- Active Comparator 3 (Active Comparator): HGP0608
  Interventions: Drug: Losartan; Drug: Placebo
- Placebo Comparator (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HCP1803 — HCP1803
  Arms: Experimental 1; Experimental 2; Experimental 3
Drug: Amlodipine — Amlodipine
  Arms: Active Comparator 1; Active Comparator 2
Drug: Losartan — Losartan
  Arms: Active Comparator 3
Drug: Placebo — Placebo
  Arms: Active Comparator 2; Active Comparator 3; Experimental 1; Experimental 2; Experimental 3; Placebo Comparator

SUMMARY:
A multicenter, randomized, double-blind, parallel, phase 2 study to assess dose-response relationship of HCP1803 in patients with essential hypertension

ELIGIBILITY:
Inclusion Criteria:

* Patient with essential hypertension who meet 140 mmHg ≤ mean sitSBP < 180 mmHg and mean sitDBP < 110 mmHg at Visit 1, Visit 2

Exclusion Criteria:

* Patient with differences between arms greater than 20 mmHg for mean sitSBP or 10 mmHg for mean sitDBP at Visit 1
* Patient with difference of ≥ 15 mmHg in mean sitSBP between Visit 1 and Visit 2
* Patient with mean sitSBP ≥ 180 mmHg or mean sitDBP ≥ 110 mmHg at Visit 1, Visit 2
* Patient with secondary hypertension

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline in sitting systolic blood pressure | baseline, 8 weeks

SECONDARY OUTCOMES:
Change from baseline in sitting systolic blood pressure | baseline, 4 weeks
Change from baseline in sitting distolic blood pressure | baseline, 4 weeks, 8 weeks
Proportion of subjects achieving blood pressure control | 4 weeks, 8 weeks
  sitSBP/sitDBP < 140/90 mmHg
Proportion of responder | baseline, 4 weeks, 8 weeks
  Change from baseline in sitSBP/sitDBP ≥ 20/10 mmHg
Change from baseline in pulse pressure(sitSBP - sitDBP) | baseline, 4 weeks, 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Moo-Yong Rhee, M.D., Ph.D., Principal Investigator — Donggguk University Ilsan Hospital
Locations (1):
- Donggguk University Ilsan Hospital, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hong SJ, Sung KC, Lim SW, Kim SY, Kim W, Shin J, Park S, Kim HY, Rhee MY; HM_APOLLO Investigators. Low-Dose Triple Antihypertensive Combination Therapy in Patients with Hypertension: A Randomized, Double-Blind, Phase II Study. Drug Des Devel Ther. 2020 Dec 31;14:5735-5746. doi: 10.2147/DDDT.S286586. eCollection 2020. PMID 33408462